CLINICAL TRIAL: NCT06639308
Title: Eendoscopic Versus Open Flexor Hallucis Longus Transfer in Managing Various Tendon Achilles Disorders
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, muhammad kamel muhammad sayed, Asisstant lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB 04-2024-100267
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Tendon Tear; Tendinopathy; Achilles Tendon Ruptures; Achilles Injuries Tendon; Achilles Tendon Surgery; Achilles Tendinopathy; Achilles Tendon Repairs/reconstructions; Haglund's Deformity
Keywords: achilles tendon rapture; achilles tendinopathy; achilles tendon transfer; fhl tendon transfer; Flexor hallucis longus tendon transfer; Haglund syndrome; endoscopic FHL transfer
MeSH Terms: conditions — Tendinopathy

STUDY DESIGN:
Intervention Model Description: •This is a Prospective, randomized control trial. The study will be conducted on 30 patients complaining of chronic Achilles tendon rupture, Achilles insertional tendinopathy, Haglund syndrome planned for FHL transfer in Assiut university hospital.
  Patients will be randomized to two groups one group endoscopic FHL will be conducted in other hand second group open FHL will be conducted.
Who Masked: Investigator, Outcomes Assessor
Masking Description: anesthesia ,
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A : open fhl tendon transfer (Active Comparator): the open surgery group The FHL tendon can be approached through the posterior longitudinal incision The FHL is confirmed by digital retraction of the tendon, watching for flexion of the hallux. Dissection of the FHL tendon is followed to the posterior talus and FHL tunnel, remaining lateral to avoid the neurovascular bundle. Release of the fibro-osseous tunnel along the posterior talus is necessary to gain length. With the hallux and ankle plantar flexed, the FHL tendon is transected as distally as possible. The tendon is fixed to the calcaneus just anterior to the Achilles stump insertion by an interference screw.
  Interventions: Procedure: Open Flexor Hallucis longus transfer to tendon achilles
- Group B : endoscopic open fhl tendon transfer (Active Comparator): • Endoscopic FHL tendon transfer: The endoscopic FHL tendon transfer is usually performed with the scope introduced through the posterolateral portal and instruments through the posteromedial portal. The FHL tendon must be identified during hindfoot working area creation. The FHL tendon is the main hindfoot endoscopic landmark as the neurovascular tibial bundle is located medial to it. First, the calcaneoplasty is completed as described. Next, the FHL tendon is harvested. The posterior fibulo-talocalcaneal ligament complex or Rouvière and Canela ligament is cut as proximal as possible in order to allow free movement of the FHL tendon and allows a straight FHL tendon trajectory to the most posterior aspect of the calcaneal bone.
  The FHL tendon is pierced with a suture passer, and a lasso loop type suture is tied to provide traction on the tendon. The foot is held in plantar flexion with the hallux flexed, relaxing the flexor hallucis longus (FHL), and the traction suture is grasped an
  Interventions: Procedure: Endoscopic Flexor Hallucis longus tendon transfer to tendon achilles

INTERVENTIONS:
Procedure: Endoscopic Flexor Hallucis longus tendon transfer to tendon achilles — The endoscopic FHL tendon transfer is usually performed with the scope introduced through the posterolateral portal and instruments through the posteromedial portal. The FHL tendon must be identified during hindfoot working area creation. First, the calcaneoplasty is completed as described. Next, the FHL tendon is harvested. A tunnel was created into calcenous the tendon is introduced into the tunnel and the tendon is secured with an interference screw of same size than the tunnel
  Other Names: Endoscopic FHL tendon transfer to tendon achilles
  Arms: Group B : endoscopic open fhl tendon transfer
Procedure: Open Flexor Hallucis longus transfer to tendon achilles — The FHL tendon can be approached through the posterior longitudinal incision The FHL is confirmed by digital retraction of the tendon, watching for flexion of the hallux. Dissection of the FHL tendon is followed to the posterior talus and FHL tunnel, remaining lateral to avoid the neurovascular bundle. Release of the fibro-osseous tunnel along the posterior talus is necessary to gain length. With the hallux and ankle plantar flexed, the FHL tendon is transected as distally as possible. The tendon is fixed to the calcaneus just anterior to the Achilles stump insertion by an interference screw.
  Other Names: Open FHL transfer to tendon achilles
  Arms: Group A : open fhl tendon transfer

SUMMARY:
* A well-established protocol for the treatment or augmentation a wide range of Achilles disorders including chronic Achilles tendon (AT) rupture, Achilles insertional tendinopathy, Haglund syndrome and among others, is a Flexor hallucis longus (FHL) tendon transfer (1-4).
* Long incisions are required for open surgical procedures, which increase the risk of skin breakdown and wound infection. These factors have contributed to the increased use of endoscopy in the surgical treatment of different Achilles pathologies. Compared to open methods, endoscopic techniques provided the advantage of managing pathology with a low risk of soft-tissue complications(4-7).
* It has been recommended to use an FHL transfer. (8-10) Its anatomic proximity prevents iatrogenic lesions of the neurovascular bundle, it fires in phase with the gastrocnemius-soleus complex, it is a stronger plantar flexor, and its axis of contractile force more closely looks similar to that of the AT. It is plantar flexion strength reinforcement, which is almost always compromised with fascial advancement alone(11). Regarding the nature of the AT's vascularization, the FHL muscle belly reaches distally into its avascular zone, which allows the repaired AT to be recruitment of an increased blood supply. Moreover, by moving muscles that perform the same function, FHL transfer preserves the ankle's natural muscular balance. (8) A recent study using magnetic resonance imaging evaluation revealed that in 60% of patients, the FHL tendon had fully integrated, and in 80% of patients, there was hypertrophy of the tendon above 15%.
* This study tends to compare the outcomes of both open and endoscopic FHL transfer in different parameters like functional outcome, wound complication, and accelerated rehabilitation.
* This is a Prospective, randomized control trial. The study will be conducted on 30 patients complaining of chronic Achilles tendon rupture, Achilles insertional tendinopathy, Haglund syndrome planned for FHL transfer in Assiut university hospital. Patients will be randomized to two groups one group endoscopic FHL will be conducted in other hand second group open FHL will be conducted.

The PICOT algorithm was preliminarily pointed out:

* P (Problem): Different Achilles disorders such as chronic Achilles tendon (AT) rupture, Achilles insertional tendinopathy, Haglund syndrome and among others.
* I (Intervention): Endoscopic FHL Transfer.
* C (Comparison): open FHL tendon transfers.
* O (Outcomes): Clinical outcomes, complications, and return to sport.
* T (Timing): ≥6 months of follow-up.

Preoperative assessment:

A- Detailed history and examination:

* Detailed history for patient complains and previous trauma or surgery.
* Physical examination for FHL, AT, any foot and ankle deformities, functional Achilles pathology or ankle range-of-motion deficits.
* VAS score, Achilles tendon Total Rupture Score - ATRS, American Orthopaedic Foot & Ankle Society (AOFAS) hindfoot score and ankle plantarflexion strength will be assessed preoperatively and at the latest follow-up (minimum of 1 year after the procedure).

Research outcome measures:

a. Primary (main): Functional outcome of endoscopic versus open FHL transfer in various TA pathology (American Orthopaedic Foot & Ankle Society (AOFAS) ankle-hindfoot score), Achilles tendon Total Rupture Score - ATRS, ankle plantarflexion strength.

.Secondary (subsidiary):

* Wound complication, skin dehiscence and infection rate.
* Expected time to complete return to sports activities or return to previous levels of activity.
* Accelerated rehabilitation.

DETAILED DESCRIPTION:
It is research that will be applied on patients with tendon Achilles disorders and planned for a Flexor hallucis longus (FHL) tendon transfer to augment and strength planter flexion power of ankle. Using endoscopic techniques provided the advantage of managing pathology with a low risk of soft-tissue complications and improve outcome.

The study will be approved from Ethical and research committee of the faculty of medicine Asyut University.

Type of the study: This is a Prospective, randomized control trial.

* Study Setting: Department of Orthopaedic and trauma surgery, Assiut university.
* Study subjects:

  1. Inclusion criteria:
  2. Chronic T.A ruptures more than 6 weeks.
  3. Non-insertional TA tendinopathy with an injury greater than 50%.
  4. Haglund deformity plus insertional Achilles tendinopathy (IAT).
  5. Patients with major degenerative tendon tissues with acute Achilles tendon rupture.
  6. Acute Achilles tendon rupture in athletic patients.
  7. Failed conservative or operatively treated ruptures healed T.A with both reduced function and significantly lengthening of the Achilles tendon after focused physiotherapy (treatment has failed to restore function to a level evaluated as satisfactory by the patients).

  b. Exclusion criteria: h. Malalignment, or end-stage tibiotalar and subtalar joint osteoarthritis. i. The presence of FHL tendon pathology. j. Acute or chronic infection. k. Sever bone loss or defects. Systemic immunodeficiency or chemotherapy c. Sample Size Calculation:

Sample size:

Based on determining the main outcome variable, the estimated minimum required sample size is 24 patients (12 patient in each group)(4)

The sample was calculated using G*power software 3.1.9.2., based on the following assumptions:

Main outcome variable is the difference between mean value of strength of planter flexion of ankle joint using the American ankle and foot functional score (AOFAS).

Based on clinical experience we expected to find large effect size difference (4)between 2 groups Main statistical test is independent t-test to detect the difference between the 2 groups.

Alpha = 0.05 Power = 0.80 Effect size = 1.2

Preoperative assessment:

A- Detailed history and examination:

* Detailed history for patient complains and previous trauma or surgery.
* Physical examination for FHL, AT, any foot and ankle deformities, functional Achilles pathology or ankle range-of-motion deficits.
* VAS score, Achilles tendon Total Rupture Score - ATRS, American Orthopaedic Foot & Ankle Society (AOFAS) hindfoot score and ankle plantarflexion strength will be assessed preoperatively and at the latest follow-up (minimum of 1 year after the procedure).

B- Radiological assessment

* Plane X-ray for ankle and foot (AP -Lateral - standing AP)
* MRI showing FHL, TA pathology and other foot or ankle pathology.

C- Surgical procedure

A-Endoscopic FHL tendon transfer:

* Patients will place in a prone position under spinal or general anaesthesia with a thigh tourniquet. Hindfoot endoscopic portals (posteromedial and posterolateral) will be located at the same level of the fibular tip or slightly distal at both sides of the Achilles tendon (with the aim to better vision and access to the insertional area of the Achilles tendon, modified portals will be located slightly distal and anterior to the classical hindfoot endoscopic portals). The posterolateral portal was used as the visualization portal and the posteromedial portal as the working portal. A distal midline Achilles portal has been described and used for Haglund resection and introduction of bioabsorbable screw may be used in some cases.
* A standardized endoscopic technique will be performed. A working area will be created when posterior soft tissue is debrided. Anatomical structures of the posterior ankle should be identified. The posterolateral aspect of the subtalar joint is first identified. Next, the scope and instruments will be redirected to the posterior area. With the shaver in contact with the superior area of the calcaneus, removal of the soft tissue and bursectomy is performed until the posterior calcaneal tubercle is visualized.
* After calcaneal bursectomy, and with the ankle in plantarflexion the anterior surface of the AT and its insertional area could be observed.
* Endoscopic calcaneoplasty: Haglund deformity can be resected with the instruments inserted through the posterolateral and posteromedial classic or modified hindfoot endoscopic portals. The calcaneal ostectomy will be performed with the burr inserted through a distal midline Achilles portal. Care should be taken to protect the AT. The cutting end of the instrument should be directed toward the bone and away from the tendon. Bone resection could be underestimated when endoscopically performed. Radiological control is recommended to observe calcaneal ostectomy. A Kirschner wire (K-wire) placed under radiological control can be used as a guide for the bone resection. If any pathology of the tendon such as intra-tendinous calcification or insertional partial tendon tear is observed, debridement of the pathological tissue can be performed with arthroscopic shaver.
* Endoscopic FHL tendon transfer: The endoscopic FHL tendon transfer is usually performed with the scope introduced through the posterolateral portal and instruments through the posteromedial portal. The FHL tendon must be identified during hindfoot working area creation. The FHL tendon is the main hindfoot endoscopic landmark as the neurovascular tibial bundle is located medial to it. First, the calcaneoplasty is completed as described. Next, the FHL tendon is harvested. The posterior fibulo-talocalcaneal ligament complex or Rouvière and Canela ligament is cut as proximal as possible in order to allow free movement of the FHL tendon and allows a straight FHL tendon trajectory to the most posterior aspect of the calcaneal bone.

The FHL tendon is pierced with a suture passer, and a lasso loop type suture is tied to provide traction on the tendon. The foot is held in plantar flexion with the hallux flexed, relaxing the flexor hallucis longus (FHL), and the traction suture is grasped and gently pulled, allowing for as distal a tenotomy as possible. Tenotomy is performed with arthroscopic scissors while the foot is maintained in the aforementioned position(9) (12).

• Once the tendon is cut, it is pulled out through the posteromedial portal. The tendon is grasped with a Krackow suture. A high-resistance suture (#0 or #2) is recommended. Then, the FHL tendon has to be introduced into a calcaneal tunnel and secured with a screw. A half-tunnel is drilled in the most posterior and superior part of the calcaneus, as close as possible to the AT. A K-wire with an eyelet introduced through the posteromedial portal is used as guide for the drill. Drilling direction should be from dorsal to plantar and centred at midpoint between medial to lateral. The diameter of the tunnel depends on the measure of the FHL tendon diameter, while the tunnel depth is at least 10 mm to 15 mm longer than the FHL tendon length obtained. Once the tunnel is drilled, suture is introduced into the eyelet of the K-wire. By pushing out the K-wire from the plantar aspect, the sutures are passed through the tunnel, and by pulling the sutures, the tendon is introduced into the tunnel. If necessary, the introduction of the FHL tendon into the tunnel can be helped with a probe. Under direct endoscopic vision, a nitinol wire is introduced into the tunnel through the posteromedial portal. Finally, with the ankle in plantarflexion the sutures are pulled to tight the FHL tendon and the tendon is secured with an interference screw of same size than the tunnel. Advancement of the screw and a final endoscopic control is performed. Incisions will be closed, and a walker boot will be applied with heel wedge in order to keep 15◦ to 20◦ of plantarflexion.

B- Open FHL transfer:

The FHL tendon can be approached through the posterior longitudinal incision The FHL is confirmed by digital retraction of the tendon, watching for flexion of the hallux. Dissection of the FHL tendon is followed to the posterior talus and FHL tunnel, remaining lateral to avoid the neurovascular bundle. Release of the fibro-osseous tunnel along the posterior talus is necessary to gain length. With the hallux and ankle plantar flexed, the FHL tendon is transected as distally as possible. The tendon is fixed to the calcaneus just anterior to the Achilles stump insertion by an interference screw.

ELIGIBILITY:
Inclusion Criteria:

* Chronic T.A ruptures more than 6 weeks.
* Non-insertional TA tendinopathy with an injury greater than 50%.
* Haglund deformity plus insertional Achilles tendinopathy (IAT).
* Patients with major degenerative tendon tissues with acute Achilles tendon rupture.
* Acute Achilles tendon rupture in athletic patients.
* Failed conservative or operatively treated ruptures healed T.A with both reduced function and significantly lengthening of the Achilles tendon after focused physiotherapy (treatment has failed to restore function to a level evaluated as satisfactory by the patients).

Exclusion Criteria:

* h. Malalignment, or end-stage tibiotalar and subtalar joint osteoarthritis. i. The presence of FHL tendon pathology. j. Acute or chronic infection. k. Sever bone loss or defects. Systemic immunodeficiency or chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-04-04 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Functional outcome of Ankle joint | one year follow up
  Functional outcome of endoscopic versus open FHL transfer in various TA pathology (American Orthopaedic Foot & Ankle Society (AOFAS) ankle-hindfoot score), ankle plantarflexion strength.

SECONDARY OUTCOMES:
Complications | one year follow up
  Wound complication( skin dehiscence and infection rate)
TIme to return to previous activity | one year follow up
  Expected time to complete return to sports activities or return to previous levels of activity.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university hospital , orthopaedic and trauma surgery department arthroscopic unit, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Attia AK, Mahmoud K, d'Hooghe P, Bariteau J, Labib SA, Myerson MS. Outcomes and Complications of Open Versus Minimally Invasive Repair of Acute Achilles Tendon Ruptures: A Systematic Review and Meta-analysis of Randomized Controlled Trials. Am J Sports Med. 2023 Mar;51(3):825-836. doi: 10.1177/03635465211053619. Epub 2021 Dec 15. PMID 34908499
- [Background] Alhaug OK, Berdal G, Husebye EE, Hvaal K. Flexor hallucis longus tendon transfer for chronic Achilles tendon rupture. A retrospective study. Foot Ankle Surg. 2019 Oct;25(5):630-635. doi: 10.1016/j.fas.2018.07.002. Epub 2018 Jul 18. PMID 30321934
- [Background] Wegrzyn J, Luciani JF, Philippot R, Brunet-Guedj E, Moyen B, Besse JL. Chronic Achilles tendon rupture reconstruction using a modified flexor hallucis longus transfer. Int Orthop. 2010 Dec;34(8):1187-92. doi: 10.1007/s00264-009-0859-1. Epub 2009 Aug 21. PMID 19697026
- [Background] Goncalves S, Caetano R, Corte-Real N. Salvage Flexor Hallucis Longus Transfer for a Failed Achilles Repair: Endoscopic Technique. Arthrosc Tech. 2015 Sep 7;4(5):e411-6. doi: 10.1016/j.eats.2015.03.017. eCollection 2015 Oct. PMID 26697296
- [Background] Hahn F, Meyer P, Maiwald C, Zanetti M, Vienne P. Treatment of chronic achilles tendinopathy and ruptures with flexor hallucis tendon transfer: clinical outcome and MRI findings. Foot Ankle Int. 2008 Aug;29(8):794-802. doi: 10.3113/FAI.2008.0794. PMID 18752777
- [Background] DeCarbo WT, Hyer CF. Interference screw fixation for flexor hallucis longus tendon transfer for chronic Achilles tendonopathy. J Foot Ankle Surg. 2008 Jan-Feb;47(1):69-72. doi: 10.1053/j.jfas.2007.09.001. Epub 2007 Nov 26. PMID 18156070
- [Background] Lee KB, Park YH, Yoon TR, Chung JY. Reconstruction of neglected Achilles tendon rupture using the flexor hallucis tendon. Knee Surg Sports Traumatol Arthrosc. 2009 Mar;17(3):316-20. doi: 10.1007/s00167-008-0693-9. Epub 2008 Dec 16. PMID 19083203
- See also: Endoscopic Flexor Hallucis Longus Transfer for Chronic Noninsertional Achilles Tendon Rupture — https://pubmed.ncbi.nlm.nih.gov/30124070/
- See also: Flexor hallucis longus tendon transfer for chronic Achilles tendon rupture. A retrospective study — https://pubmed.ncbi.nlm.nih.gov/30321934/